CLINICAL TRIAL: NCT03771638
Title: DOT Diary Longitudinal Pilot: A Mobile App for Pre-Exposure Prophylaxis Adherence in Young Men
Brief Title: DOT Diary Mobile App for Pre-Exposure Prophylaxis Adherence in Young Men
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Public Health Foundation Enterprises, Inc. (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); San Francisco Department of Public Health (Other Government); Emory University (Other); AiCure (Industry)
Responsible Party: Principal Investigator, Susan Buchbinder, Director, Bridge HIV, Public Health Foundation Enterprises, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-25821; 1R01MH109320-01 (NIH)
Record Dates: First submitted 2018-12-03; First posted 2018-12-11 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Adherence, Medication; Risk Behavior; Pre-Exposure Prophylaxis; HIV Prevention
Keywords: Adherence; PrEP; HIV Prevention; Truvada; HIV Risk Reduction; Mobile App
MeSH Terms: conditions — Medication Adherence; Risk-Taking | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: Randomized, controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- DOT Diary Intervention (Experimental): DOT Diary mobile app and Emtricitabine / Tenofovir Disoproxil Oral Tablet (once daily)
  Interventions: Drug: Emtricitabine / Tenofovir Disoproxil Oral Tablet; Other: DOT Diary mobile app
- DOT Diary Control (Other): Standard of care for Emtricitabine / Tenofovir Disoproxil Oral Tablet (once daily)
  Interventions: Drug: Emtricitabine / Tenofovir Disoproxil Oral Tablet

INTERVENTIONS:
Drug: Emtricitabine / Tenofovir Disoproxil Oral Tablet — Open label daily emtricitabine/tenofovir disoproxil oral tablet
  Other Names: Truvada
Other: DOT Diary mobile app — DOT Diary mobile application for tracking medication adherence and sexual activities.
  Arms: DOT Diary Intervention

SUMMARY:
The researchers are working with a technology company, AiCure, to develop a smartphone app, DOT Diary, which combines two drug adherence strategies. DOT Diary reminds people when it is time to take their medication, and uses motion-sensing technology to visually and automatically confirm the pill was swallowed. The goal of this study is to assess the impact of the app on adherence to HIV pre-exposure prophylaxis (PrEP) for the prevention of HIV.

DETAILED DESCRIPTION:
In the DOT Diary research project, the AiCure automated directly observed therapy (aDOT) smartphone app has been adapted for use in monitoring and supporting HIV pre-exposure prophylaxis (PrEP) use among young men who have sex with men (YMSM). The aDOT app uses automated directly observed therapy (DOT) that use the smartphone camera and artificial intelligence software to confirm that the right person is taking the right medication at the right time. A sexual diary has been integrated into the aDOT app to assist YMSM in understanding whether they are receiving protection from PrEP for individual sexual episodes, and when it is particularly important to take PrEP (e.g. after a sexual episode). Specifically, the sexual diary allows participants to track sexual encounters, sexual behaviors that occurred in each encounter, and rating characteristics of partners. The app provides a calendar displaying all days in which PrEP medication was taken, and all days in which sexual activity occurred, allowing participants to see coverage of sexual encounters with PrEP. Based on pharmacokinetic and pharmacodynamic data from prior PrEP trials, the app will also indicate the estimated level of protection achieved from PrEP (e.g. low, medium, high), and also provide personalized messages on the additional numbers of doses needed to maximize protection.

In the next stage of app development and assessment, the researchers will conduct the DOT Diary Longitudinal Pilot to assess the impact of the app on PrEP adherence as measured by pharmacokinetic measures of PrEP use (tenofovir diphosphate [TFV-DP] and emtricitabine triphosphate [FTC-TP] levels in dried blood spots [DBS]). The researchers will also assess the concordance of TFV-DP and FTC-TP in DBS with adherence measured by DOT Diary, and the acceptability and ease of use of the app over a longer (24-week) period. This pilot study will allow evaluation and further refinement of the app in preparation for testing in a larger efficacy trial among YMSM at risk for HIV acquisition. The researchers will conduct this pilot protocol among YMSM in Atlanta and San Francisco Bay Area, two metropolitan regions heavily impacted by HIV, yet differing in sociodemographics, as well as in the availability and uptake of HIV prevention services, including PrEP. These diverse research locations will allow collection of data to inform app development among a broad group of YMSM.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as a man
* Age 18-35 at enrollment
* Reports having insertive or receptive anal sex with a man or trans woman in the past 12 months and one or more of the following criteria in the last 12 months:

  * Any condomless anal sex outside of a mutually monogamous relationship with an HIV-negative partner
  * Two or more anal sex partners
  * Self-reported sexually transmitted infection (STI; gonorrhea, chlamydia, syphilis)
  * Having a known HIV-positive sexual partner
* HIV-negative as determined by a negative 4th generation HIV test at screening and negative rapid 4th generation test at enrollment
* Willing to initiate PrEP
* Eligible to take PrEP

  * Creatinine clearance ≥60 ml/min as estimated by Cockcroft-Gault equation at screening
  * Hepatitis B surface antigen (HBsAg) negative
* Willing and able to provide written informed consent
* Able to read and speak English
* Smartphone ownership compatible with DOT Diary app
* Meets local locator requirements
* Lives, works or plays in Atlanta Metropolitan Area, San Francisco, Alameda, Marin, Contra Costa, Santa Clara, or San Mateo Counties

Exclusion Criteria:

* PrEP use within the past 4 months (PrEP naive participants will be prioritized)
* Any reactive HIV test at screening or enrollment
* Signs or symptoms of acute HIV infection at screening or enrollment
* History of pathological bone fracture not related to trauma
* Taking nephrotoxic medications
* History of participation in the active arm of an HIV vaccine trial
* In a mutually monogamous sexual relationship with an HIV-negative partner for the past 12 months
* Unable to commit to study participation for 24 weeks
* Any medical, psychiatric, or social condition or other responsibilities that, in the judgment of the investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-identify as a man
Enrollment: 100 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Buchbinder, MD, Principal Investigator — Bridge HIV, San Francisco Department of Public Health
Locations (2):
- United States (2):
  - Bridge HIV, San Francisco Department of Public Health, San Francisco, California
  - Emory University, School of Public Health, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Velloza J, Liu AY, Katz AWK, van der Straten A, Siegler AJ, Scott H, Wilde G, Lockard A, Christie RH, Buchbinder SP. Acceptability of an automated directly observed therapy (DOT) application for PrEP adherence support among young men who have sex with men: a qualitative exploration. AIDS Care. 2024 Nov;36(11):1704-1718. doi: 10.1080/09540121.2024.2397133. Epub 2024 Sep 2. PMID 39222964

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited into the study using online recruitment techniques and outreach into venues frequented by men who have sex with men. The protocol opened on February 1, 2019 and study follow-up was complete on April 21, 2020. Participants were recruited from the Atlanta Metropolitan Area or the greater San Francisco Bay Area, with 50 participants recruited from each location.
Pre-assignment Details: Participants were screened for behavioral and medical eligibility. If they met study eligibility criteria and were willing to consent to participate, they were enrolled in the study.
Period: Overall Study
Arm/Group | DOT Diary Intervention | DOT Diary Control
Started | 66 | 34
Completed | 60 | 29
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Population: This is a cohort of HIV uninfected men who have sex with men who qualify for taking HIV pre-exposure prophylaxis.
Groups:
- Total: Total of all reporting groups
Arm/Group | DOT Diary Intervention | DOT Diary Control | Total
Number analyzed (Participants) | 66 | 34 | 100
Age, Continuous [Mean (Full Range); unit: years] | 26.0 [18 to 35] | 25.9 [18 to 35] | 26 [18 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 66 | 34 | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants could be listed as having more than one race/ethnicity
  Participants
    Asian/Pacific Islander | 10 | 4 | 14
    Black/African American | 19 | 7 | 26
    Latino | 15 | 7 | 22
    White | 21 | 15 | 36
    Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 66 | 34 | 100
Sexual orientation [Count of Participants; unit: Participants] — Data are missing for 2 participants
  Participants
    Bisexual | 5 | 6 | 11
    Gay | 56 | 27 | 83
    Queer | 3 | 1 | 4
    Missing | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Effect of DOT Diary App on PrEP Adherence
Description: Measurement of PrEP Adherence as measured by TFV-DP level >=700 fmol/punch in DBS among young MSM initiating PrEP
Time Frame: 24 weeks
Population: Participants who were retained at 24 weeks and had dried blood spot for TFV-DP levels
Measure: Count of Participants; unit: Participants
Arm/Group | DOT Diary Intervention | DOT Diary Control
Number analyzed (Participants) | 58 | 29
Participants | 39 | 19
Statistical Analysis 1: Comparison: DOT Diary Intervention vs DOT Diary Control; Null hypothesis: no difference in PrEP adherence levels between DOT Diary Intervention and Control arms; Test type: Superiority — Minimum detectable effects: Under assumptions of the adherence of DBS TFV-DP levels >=700 fmol/punch in the control condition as 60% and intraclass correlation of repeated binary measures of DBS TFV-DP of 0.69, and retention of 80% of participants at 24 weeks, we will have 80% power in 2-sided tests with a type-1 error rate of 5% to detect average between-group differences in adherence of 23 percentage points; p = 0.94, GEE Poisson models — GEE poisson models with robust standard errors were used to assess DBS adherence rates, averaged across visits; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.75 to 1.36]

2. Primary Outcome: Concordance of TFV-DP and FTC-TP in DBS With Adherence Measured by DOT Diary App
Description: As a measure of concordance between DBS measurements and aDOT-based assessments of PrEP adherence: Number of specimens with < 700 fmol/punch or >= 700 fmol/punch agreement with number of participants reporting PrEP use < 4 days/week or 4-7 days/week at weeks 6, 12, 18, 24
Time Frame: 6, 12, 18, 24 weeks
Population: DOT Diary Intervention arm with specimens collected at weeks 6, 12, 18, and 24.
Measure: Number; unit: number of measures by DBS and aDOT
Arm/Group | DOT Diary Intervention
Number analyzed (Participants) | 66
number of measures by DBS and aDOT
  specimens < 700 fmol/punch and PrEP use reported < 4 days/week | 34
  specimens < 700 fmol/punch and PrEP use reported 4-7 times/week | 29
  specimens >=700 fmol/punch and PrEP use reported < 4 days/week | 13
  specimens >= 700 fmol/punch and PrEP use reported 4-7 times/week | 135
Statistical Analysis 1: Comparison: DOT Diary Intervention; Kappa statistic to assess concordance between DBS measurement and self-reported PrEP use; Test type: Other; Kappa; Kappa statistic = 0.49, 95% CI 2-sided [0.36 to 0.62]

3. Primary Outcome: DOT Diary Mobile App Acceptability
Description: Combined descriptive analysis of key attributes of acceptability of DOT Diary over 24 weeks by YMSM on PrEP, in order to identify potential improvements to the app to maximize acceptability. This was measured using the System Usability Scale, with minmum value of 0 and maximum value of 100. This is a scale that uses a 10-item questionnaire with a 5-point Likert scale from strongly agree to strongly disagree. Scores are summed and the final score is multiplied by 2. Higher scores mean a better outcome.
Time Frame: 24 weeks
Population: Participants randomized to the DOT Diary Intervention arm who completed a system usability score measure at 24 weeks. Data are missing for 6 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DOT Diary Intervention
Number analyzed (Participants) | 60
score on a scale | 77.9 (14.7)

4. Primary Outcome: DOT Diary Mobile App Ease of Use
Description: Descriptive analysis of key attribute of ease of use of DOT Diary over 24 weeks by YMSM on PrEP. Participants were asked if the DOT Diary app was easy to use and answered using a Likert Scale from 1= Strongly disagree, 2= Disagree, 3= Neutral, 4= Agree, 5= Strongly agree. A higher score indicates a better outcome.
Time Frame: 24 weeks
Population: Participants randomized to the DOT Diary Intervention arm who completed the usability question at week 24.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | DOT Diary Intervention
Number analyzed (Participants) | 60
score on a scale | 4.3 [1 to 5]

5. Secondary Outcome: PrEP Coverage of Sexual Acts (Prevention-effectiveness Adherence) as Measured by DOT Diary
Description: Percentage of total anal sex acts across the 30 participants covered by use of PrEP for 4-7 days prior to that sex act, as measured by a-DOT. This is only for the a-DOT arm of the study.
Time Frame: 6, 12, 18, 24 weeks
Population: Participants in the DOT Diary group who reported anal sex in their diary.
Measure: Number; unit: % ot 100 sex acts covered by PrEP
Units Other Than Participants: sex acts covered by PrEP
Arm/Group | DOT Diary Intervention
Number analyzed (Participants) | 30
Number analyzed (sex acts covered by PrEP) | 100
% ot 100 sex acts covered by PrEP | 93

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Standard definitions for AE and SAE apply
Groups:
- DOT Diary Intervention Arm: This is the arm that was randomized to receive the DOT Diary intervention
- DOT Diary Control Arm: This is the arm that was randomized to receive the standard of prevention.
Arm/Group | DOT Diary Intervention Arm | DOT Diary Control Arm
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/34
Other Adverse Events (participants affected / at risk) | 0/66 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT03771638/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT03771638/SAP_002.pdf